CLINICAL TRIAL: NCT04960904
Title: Study Evaluating the Performance and Safety in the Medium and Long Term of Implant-prosthetic Systems Including Ranges of Dental Implants and Prosthetic Components Global D: In-Kone® U,In-Kone® P,twinKon®,EVL® S,EVL® K,EVL® C
Brief Title: Study Evaluating the Performance and Safety in the Medium and Long Term of Global D Implant-prosthetic Systems
Status: Recruiting | Type: Observational
Sponsor: Global D (Industry)
Responsible Party: Sponsor
Other Study IDs: 1905-G-IMP-DENT-R
Record Dates: First submitted 2021-06-30; First posted 2021-07-14 (Actual); Last update posted 2025-04-02 (Actual); Status verified 2025-03

CONDITIONS: Dental Implants
Keywords: dental implant; survival rate; performance

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (6):
- In-Kone® UNIVERSAL: Implant-prosthetic systems made with dental implants and prosthetic components of the ranges In-Kone® UNIVERSAL, including the former 3.0 range now named In-Kone® Universal NR (narrow), and including the In-Kone® Universal WD (wide).
  Interventions: Device: Dental implant surgery with implants
- In-Kone® PRIMO: Implant-prosthetic systems made with dental implants and prosthetic components of the ranges In-Kone® PRIMO
  Interventions: Device: Dental implant surgery with implants
- twinKon®: Implant-prosthetic systems made with dental implants and prosthetic components of the ranges twinKon®
  Interventions: Device: Dental implant surgery with implants
- EVL® S: Implant-prosthetic systems made with dental implants and prosthetic components of the ranges EVL® S
  Interventions: Device: Dental implant surgery with implants
- EVL® K: Implant-prosthetic systems made with dental implants and prosthetic components of the ranges EVL® K
  Interventions: Device: Dental implant surgery with implants
- EVL® C: Implant-prosthetic systems made with dental implants and prosthetic components of the ranges EVL® C
  Interventions: Device: Dental implant surgery with implants

INTERVENTIONS:
Device: Dental implant surgery with implants — Adult patients who have had dental implant surgery.

SUMMARY:
This study is set up within the framework of the European Union regulation 2017/745 on medical devices. Its objective is to confirm the performance and safety in the medium and long term of implant-prosthetic systems including Global D dental implants: In-Kone® UNIVERSAL, In-Kone® PRIMO, twinKon®, EVL® S, EVL® K and EVL® C.

DETAILED DESCRIPTION:
Study design: Ambispective multi-center observational study, on a single patient group per implant, constituting a consecutive and exhaustive series of subjects, without selection.

Investigators:Twelve centers participated to the study in France and one in Greece.

The objectives are evaluate the 5-year follow-up performance and safety of Global D dental implant ranges, which consist of collecting data at a 5-year follow-up visit (prospectively or retrospectively). All previous data is collected retrospectively from the patient's file. The study has been extended to 7/8 years and up to 10 years follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Male or female
* Major (s) at the time of the implantation
* Having needed implant surgery with one or more Global D devices:
* between October 1, 2013 - June 30, 2015 for EVL® S, EVL® K and EVL® C, In-Kone® UNIVERSAL and In-Kone® PRIMO implants
* between January 1, 2013 - June 30, 2015 for twinKon® implants
* Affiliated or benefiting from French Social Security
* Not opposing the use of their data
* Having carried out his annual follow-up visit at 5, 7/8 and 10 years or any other visit motivated by the removal of the implant during the 10 years

Exclusion Criteria:

* Patient unable to understand information related to his/her participation in the study
* Deceased patient, date of death after the date of implantation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult male or female patients who have had dental implant surgery. In the perspective of being able to obtain follow-up data at least 5 years and up to 10 years and the series to be continuous and exhaustive, the implantation period will be limited from
  * October 1, 2013 to June 30, 2015 for EVL® S, EVL® K and EVL® C, In-Kone® UNIVERSAL and In-Kone® PRIMO implants
  * January 1, 2013 to June 30, 2015 for twinKon® implants
Sampling Method: Non-Probability Sample
Enrollment: 514 (Estimated)
Dates: Start 2019-11-12 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-01-31 (Estimated)

PRIMARY OUTCOMES:
Survival rate | 5 years
  Survival rate at 5 years, 7/8 years and 10 years minimum defined by the rate of implants in situ

SECONDARY OUTCOMES:
Implant system stability | 1-4 month, 6-12 month, 5 years, 7/8 years and 10 years after surgery
  Implant system stability of all follow-up visits. Stability of the implant system is assessed by the investigator at each visit. The variable collected is YES for stable implant and NO for unstable implant.
The success rate | 5 years, 7/8 years, 10 years
  The success rate at 5 years, 7/8 years and 10 years defined by the rate of stable implants without pain or sensitivity at the implant level, with the absence of peri-implantitis and osteolysis;
Appearance of the gum | 5 years, 7/8 years, 10 years
  Appearance of the gum based on the visual appearance of the gum will be collected. Several choices are possible: Inflammation / Gingival recession / Absence of keratinized tissue band around the crown
Adverse events and complications | Up to 5 years, 7/8 years, and 10 years of follow-up
  Nature, number, severity and degree of relationship of adverse events, serious or not, reported as implant-related or unrelated for non-serious adverse events, immediate or delayed at all visits
Score of Quality of life (OHIP-14 - The Oral Health Impact Profile) | 5 years, 7/8 years, 10 years
  The score obtained from the satisfaction and quality of life questionnaire (OHIP-14) at 5 years The Oral Health Impact Profile 14 (OHIP-14) [14] is a questionnaire measuring the impact of the prosthetic restoration on the patient's well-being and quality of life. The patient answers fourteen questions grouped into seven domains (functional limitation, physical pain, psychological discomfort, physical disability, psychological disability, social disability and handicap) . For each question, the patient can answer with one of the following values: never:0, almost never:1, occasionally:2, quite often:3, very often:4. The sum of the values for each question gives a score that can vary from 0 to 56. A high score reflects a high level of discomfort.

CONTACTS AND LOCATIONS:
Overall Officials: Jean Pierre AXIOTIS, MD, Principal Investigator — Dental surgeon
Locations (2):
- Dental practice, Andrézieux-Bouthéon, France
- Dental practice, Athens, Greece

IPD SHARING:
Plan to Share IPD: No